CLINICAL TRIAL: NCT01431911
Title: Outcomes Associated With Early or Delayed Maintenance Treatment Post-Chronic Obstructive Pulmonary Disease Exacerbation
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113898
Record Dates: First submitted 2011-06-23; First posted 2011-09-12 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed with COPD: Patients diagnosed with COPD using ICD codes with a COPD-related exacerbation and receiving maintenance therapy
  Interventions: Drug: Early maintenance treatment; Drug: Delayed Maintenance treatment

INTERVENTIONS:
Drug: Early maintenance treatment — Various classes of COPD maintenance treatment initiated within 30 days post index COPD exacerbation (hospitalization/ED visit)
Drug: Delayed Maintenance treatment — Various classes of COPD maintenance treatment initiated after 30 days post index COPD exacerbation (hospitalization/ED visit)

SUMMARY:
The timing of initiating short-term treatment for COPD exacerbations with oral corticosteroids and/or antibiotic therapy has been shown to influence the recovery time of exacerbations with early initiation of exacerbation therapy having a faster symptom recovery compared to delayed initiation. While oral corticosteroids and/or antibiotic therapy are crucial for immediate exacerbation therapy, maintenance therapy with controller medications for COPD has been recommended to reduce the risk of future exacerbations. The initiation of maintenance therapy after a COPD exacerbation has been shown to be beneficial in the reduction of risk of future exacerbations. However, there is a lack of information on whether the timing of this initiation influences the risk of future exacerbations. The following study evaluates the impact of early versus delayed initiation of controller medication therapy for maintenance treatment following a COPD-related exacerbation on outcomes of future exacerbations and costs in patients with COPD.

DETAILED DESCRIPTION:
Study period for this analysis will range from January 2003 through June 2009. Patients with at least one COPD exacerbation will be selected as the initial population. Three types of COPD exacerbations will be identified: 1) hospitalization with a primary discharge diagnosis code for COPD, 2) an emergency department (ED) visit with a primary diagnosis code for COPD, 3) physician visit with a dispensing of oral corticosteroid (OCS) or antibiotic (ABX) within 5 days of the visit. Only the first two will be selected as index exacerbations, which is defined as the first chronologically occurring exacerbation for a patient. For hospitalization exacerbations the discharge date of the hospitalization will be the index date and for ED exacerbations the date of the visit will be the index date. The pre-index period will be defined as the 1-year period before index date and the post-index period will be defined as 1-year period after index date. The enrollment period will thus range from January 1, 2004 through June 30, 2008. The post-index period will be used to identify the date of receipt of prescription for first COPD maintenance medication. This date of receipt will be used to compute the time to start maintenance treatment. Maintenance treatment refers to the use of controller medications.

Specifically the study hypothesis for the primary outcome being tested was:

Ho: There is no difference in risk of COPD-related hospitalization/ED visit between early and delayed cohorts Ha: There is a difference in risk of COPD-related hospitalization/ED visit between early and delayed cohorts

Hypothesis for the key secondary outcome of COPD-related costs that was tested was:

Ho: There is no difference in COPD-related costs between early and delayed cohorts Ha: There is a difference in COPD-related costs between early and delayed cohorts

ELIGIBILITY:
Inclusion Criteria:

* at least 40 years of age,
* continuously enrolled for medical and pharmacy benefits during their pre- and post-period
* diagnosis of COPD (ICD 491.xx, 492.xx, 496.xx)

Exclusion Criteria:

* Patients were excluded if they had MTx in the pre-index period (to ensure inclusion of MTx-naïve patients) or if they received their first MTx during 181 to 365 days of the post-period (as dispensing of MTx unlikely to be related to the index exacerbation).
* Additionally, patients were excluded if they had any of the following comorbid conditions anytime during the study period: respiratory cancer, cystic fibrosis, fibrosis due to, bronchiectasis, pneumonociosis, pulmonary fibrosis, pulmonary tuberculosis, or sarcoidosis, and
* also if they had other doses (unapproved in the US) of fluticasone propionate-salmeterol xinafoate combination (100/50 mcg or 500/50 mcg) or budesonide dipropionate-formoterol fumarate fixed dose combination (any dose).

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients meeting study criteria mentioned belowwere classified into two cohorts, early and delayed, based on timing of (maintenance treatment) MTx after the index date - 0 to 30 days and 31 to 180 days, respectively. A 30-day period was chosen to define early initiation based on sample size considerations and recent evidence demonstrating the increased risk of subsequent exacerbations during an 8-week period following an initial exacerbation [Hurst JR 2009]. Outcomes were computed for and compared between these two cohorts. An incremental analysis evaluating the effect of delaying MTx by every 30 days was also done classifying patients into six categories based on 30-day increments of starting MTx (0 to 30 days, 31 to 60 days, 61 to 90 days, 91 to 120 days, 121 to 150 days, and 151 to 180 days) (Figure 1). Outcomes were then compared across the 6 categories thereby allowing assessment for every 30-day increment up to 180 days after the index date.
Sampling Method: Non-Probability Sample
Enrollment: 3806 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
COPD hospitalization/ED visit | Up to 6 years (January 1, 2003 through June 30, 2009)
  Risk and number of COPD exacerbations will be computed in the post-index period. Hospitalization with a primary discharge diagnosis code (ICD code 491.xx, 492.xx, and 496.xx) for COPD. ED visit will be defined as COPD related if accompanied by diagnosis code for COPD.

SECONDARY OUTCOMES:
COPD-related ED visit | Up to 6 years (January 1, 2003 through June 30, 2009)
  The risk and proportion of patients with a COPD-related exacerbation requiring ED visit was defined as a COPD-related ED visit.
COPD-related hospitalization | Up to 6 years (January 1, 2003 through June 30, 2009)
  risk and number of COPD hospitalizations will be computed in the post-index period. Hospitalization with a primary discharge diagnosis code (ICD code 491.xx, 492.xx, and 496.xx) for COPD will be captured.
COPD-related Phy+Rx visit | January 1, 2003 through June 30, 2009 (up to 6 years)
  Risk and number of COPD-related physician office visit with a dispensing for oral corticosteroid (OCS) or antibiotic (ABX) within 5 days of the visit
COPD related Costs | January 1, 2003 through June 30, 2009 (up to 6 years)
  COPD related medical, pharmacy and total costs. Costs were standardized to 2009 US dollars (USD) using consumer price index for US medical care.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline